CLINICAL TRIAL: NCT01737658
Title: Insulin Resistance and Cognitive Dysfunction in Obese Adolescents: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12041
Record Dates: First submitted 2012-11-05; First posted 2012-11-29 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Program upon enrollment (Other): Subject will receive exercise intervention immediately upon enrollment to study
  Interventions: Other: Exercise Program
- Exercise Program 6 months after enrollment (Other): Subject will be enrolled into study and then receive exercise intervention 6 months after enrollment.
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Exercise Program — Exercise Program for Obese Adolescents

SUMMARY:
Obese Adolescents will be evaluated for insulin resistance and cognitive dysfunction.

DETAILED DESCRIPTION:
The short-term goal of this project is to conduct a feasibility study at Winthrop University Hospital to determine how well extremely obese (BMI > 99%tile corrected for age) children and adolescents can be recruited into an exercise program and evaluated in an efficient fashion, and to identify particular strategies (e.g., medical examination feedback) that can serve as potential benefits to research subjects and their families. In addition investigators will evaluate the effect of the exercise program on physical fitness, insulin resistance, and neurocognitive functioning as well as the relationship between insulin sensitivity and neurocognitive function among adolescents who participate in the exercise program.

The long-term goal of this project is to evaluate a large, multi-ethnic sample of adolescents, 14 to 19 years of age, to systematically assess cognitive function and school performance, fitness and examine the relationship between performance on those outcome variables and a variety of biomedical and psychosocial factors that may directly or indirectly influence brain function and test-taking performance.

High body mass index (BMI) among children and adolescents continues to be a public health concern in the United States. The most recent figures from the National Health and Nutrition Examination Survey (NHANES) for 2007-2008 report that 18.1% (95% CI, 14.5%-21.7%) of 12- through 19-year-old adolescents were at or above the 95th percentile of BMI for age. Children with high BMI often become obese adults, and obese adults are at risk for many chronic conditions. High BMI in children may also have immediate consequences, such as elevated lipid concentrations and blood pressure.

It now appears that neurocognitive dysfunction is also more common in obese children and adolescents. In a large population study of 2,519 children, 8 to 16 years of age, a brief neuropsychological assessment showed a statistically significant, albeit modest relationship between cognitive test scores and BMI that persisted after adjusting for confounding variables. Obesity is also associated with several conditions which known to affect brain function, including sleep apnea, insulin resistance, hypertension, and chronic inflammatory factors (e.g., by these variables cannot be determined, unfortunately, because those variables were not measured.

It is important to note, however, that there is not complete agreement on linkages between obesity and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subject's ages 14 to 19 years old, extremely obese (BMI ≥ 99th percentile).
* Clearance by pediatric cardiologist, including evaluation of V02Max.

Exclusion Criteria:

* Male and female less than 14years of age or more than 19 years of age.
* Patients with type 1 or type 2 diabetes
* Patients with serious medical conditions.
* Anyone who is deemed inappropriate by pediatric cardiologist during clearance evaluation.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2012-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Formal exercise intervention and cognitive dysfunction in obeses adolescents | 1 year
  To measure the feasibility of recruiting extremely obese (BMI > 99%tile corrected for age) children and adolescents into an exercise program and evaluate their physical fitness.

SECONDARY OUTCOMES:
Systemic and Cognitive effects of adding exercise program to obese adolescent's lifestyle. | 1 year
  To assess the physical fitness among participating children and adolescents before and after completion of the exercise program.
Systemic and Cognitive effects of adding exercise program to obese adolescent's lifestyle. | 1 year
  To evaluate the change in insulin sensitivity and neurocognitive function among participating children and adolescents before and after completion of the exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Siham Accacha, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States